CLINICAL TRIAL: NCT04041193
Title: An Innovative Disease-net Management Model for Non-communicable Diseases: a System for Integrated Home-care and Assisted Rehabilitation for Wellbeing
Brief Title: An Innovative Disease-net Management Model for Non-communicable Diseases (SIDERA^B)
Acronym: SIDERA^B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Università Carlo Cattaneo , Castellanza (Unknown); University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FdG_SIDERAb_01
Record Dates: First submitted 2019-06-26; First posted 2019-08-01 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease (PD); Chronic Heart Failure (CHF); Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Parkinson Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIDERA^B (Experimental): Behavioral: telerehabilitation activities Participants will receive 3months (Chronic Heart Failure) or 4 months (Chronic Obstructive Pulmonary Disease and Parkinson Disease) 5 sessions/week of an individualized telerehabilitation program at home. The sessions will initially be tailored to the patient's baseline characteristics. The exercise program will be charged by the therapist weekly. Each patient's performed session will be reviewed by the therapist.
  Interventions: Behavioral: SIDERA^B
- usual care (Active Comparator): Behavioral: paper and pencil activities as usual rehabilitation at home Participants will receive 3months (Chronic Heart Failure) or 4 months (Chronic Obstructive Pulmonary Disease and Parkinson Disease) of a usual rehabilitation program.
  Interventions: Behavioral: Usual Care Program

INTERVENTIONS:
Behavioral: SIDERA^B — The group will receive a kit home-based (a tablet home, access to a daily individualized training program). Five sessions for a week (3 components: monitoring, motor rehabilitation acitivities, motivational support)
  Arms: SIDERA^B
Behavioral: Usual Care Program — Usual Care program activities (paper and pencil at home)
  Arms: usual care

SUMMARY:
The SIDERA^B telerehabilitation system is enabled by a multi-domain, multi-device platform providing at home multi-component rehabilitation, targeting cardiovascular (Chronic Heart Failure, CHF), pulmonary (Chronic Obstructive Pulmonary Disease, COPD) and neurodegenerative (Parkinson Disease, PD) chronic diseases. The rehabilitation program embeds engagement activities for patient and caregiver, to empower appropriation of the SIDERA^B care routines and fuel their well-being resources.

The multidisciplinary layering of SIDERA^B is reflected in the validation protocol including a) clinical and well-being evaluation through a cross-over study confronting usual care with the SIDERA^B activities; b) technological evaluation: Health Technology Assessment for organizational, legal and equity impacts; c) economic evaluation: process mapping and budget impact analysis to define a sustainable reimbursement process for the innovative telerehabilitation pathway.

ELIGIBILITY:
Inclusion criteria:

1. agreement to participate, with the signature of the informed consent form.
2. availability of a caregiver/study partner, who agrees to support the participant through the SIDERA^B program.
3. living in one's own home.
4. clinical diagnosis of Chronic Heart Failure (CHF) and

   1. functional New York Heart Association (NYHA) class II and III with an Ejection Fraction (EF) ≤ 40%
   2. etiology of CHF primitive or post-ischemic.
5. clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD) and

   1. COPD diagnosis according to the American Thoracic Society (ATS) and the European Respiratory Society (ERS) criteria with FEV1/FVC ratio <70%
   2. presence of airway limitation according to ATS/ERS and GOLD criteria.
6. clinical diagnosis of Parkinson Disease (PD) and

   1. PD diagnosis according to the MDS criteria (Postuma et al., 2015)
   2. staging between 1.5 and 3 on the Hoehn & Yahr scale (Goetz et al., 2004)
7. age between 18 and 85 years.

Exclusion Criteria:

1. presence of comorbidities that may prevent you from undertaking a secure home program or determining clinical instability (i.e. severe orthopedic or severe cognitive deficits).
2. presence of risk conditions for safety under strain in patients with CHF (i.e. severe symptomatic aortic stenosis, evidence of ischemia due to minimal/low-intensity efforts).
3. COPD patients who do not need rehabilitation treatment (GOLD 1 / A class) or with severe COPD (GOLD 4 / D class)
4. COPD patients with overlap with other respiratory diseases or not in treatment or in the absence of good ventilatory compensation in the last 6 months
5. COPD with global respiratory failure with PaCO2> 55 mmHg
6. PD patients with other neurological pathologies or with severe psychiatric complications
7. pathological score to a screening test for cognitive impairment (Montreal Cognitive Assessment test - MoCA test <17.54; Conti et al., 2015).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Activation of Patients as measured by Patient Activation Measure 13 (PAM13) scale | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  Patient Activation Measure 13 (PAM13) is a 13-item scale that assesses a person's underlying knowledge, skills and confidence integral to managing his or her health and healthcare. PAM13 total score ranging from 0 to 100. Higher values represent a better outcome. Specifically, individuals in the lowest activation level do not yet understand the importance of their role in managing their health and have significant knowledge gaps and limited self-management skills. Individuals in the highest activation level are proactive with their health, have developed strong self- management skills, and are resilient in times of stress or change.
Change in activity and participation as measured by the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  WHODAS 2.0 covers six domains of functioning including Cognition, Mobility, Self-care, Getting along, Life activities, Participation. Scores assigned to each item are on a 5-point scale ranging from (0) "none" to (4) "extreme" with higher scores indicating a higher disability. The 36-item version will be administered and both summary scores (score range 0-144 with higher numbers indicating higher disability) and domain-specific scores for the six different functioning domains (score range 0-24 for each domain with higher numbers indicating higher disability) will be considered.

SECONDARY OUTCOMES:
Change in patient's self-rated health as measured by EuroQol five dimensions (5D) and five levels (5L) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The EQ-5D-5L (EQ-5D-5L, The EuroQol Group, 1990; Janssen et al.,2013) is a measure of health status that consists of the EQ-5D descriptive system and of the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A total of 3125 possible health states are defined, ranging from 1111 (no problems in all dimensions) to 5555 (extreme problems in all dimensions). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labeled 'The best health you can imagine' (scored as "100") and 'The worst health you can imagine' (scored as "0").
Change in health status scores as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ; Green et al., 2000; ad. it.: Miani et al., 2003) only in patients with Chronic Heart Failure | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status over six domains: symptoms;physical function;quality of Life; social Limitation; Self-efficacy; symptom Stability. Summary scores will be computed: the "Clinical Summary Score" including total symptom and physical function scores; the" Overall Summary Score" including the total symptom, physical function, social limitations and quality of life scores. KCCQ responses are provided along a rating scale continuum with equal spacing from worst to best.
Change in health-related quality of life as measured by Parkinsons' Disease (PD) Questionnaire (PDQ) only in PD patients | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The PDQ-39 (Jenkinson, 1997; ad. it.: Galeoto et al., 2018) is a 39-item self-administered questionnaire. It offers a patient-reported measure of health status and quality of life and is the most frequently used disease-specific health status measure and assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations, and communication. The score for each question ranges from zero (0) to four (4): "never"=0; "occasionally"=1; "sometimes"=2; "often"= 3; "always"=4. the final score is the result of the following equation: the sum of each question score divided by the result times 4 (the maximal score for each question), divided by the total number of questions. This result is multiplied times by 100. Each dimension score ranges from 0 to 100 in a linear scale, in which zero is the best and 100 the worst quality of life.
Change in health status scores as measured by St George's Respiratory Questionnaire (SGRQ) only in patients with COPD. | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  SGRQ (Jones, P. W., Quirk, F. H., & Baveystock, C. M. 1991) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. It is composed of two parts with three components: Part 1: Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall. Scaling of items is heterogenous, with Part I (Symptoms) adopting several scales and Part II (Activity and Impacts) adopting a dichotomous (true/false) scale except for last question (4-point Likert scale). Scores range from 0 to 100, with higher scores indicating more limitations.
Change in care-relationship as Measured by Mutuality Scale (MS) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The MS (Archbold et al., 1990; Pucciarelli et al., 2016; ad. it.: Dellafiore et al., 2018) is a 15-item instrument that measures mutuality in care-relationship. Each item is scored on a 5-point Likert-type scale from 0 ( not at all ) to 4 ( a great deal ). The total scale score ranges from 0 to 60: higher scores mean greater mutuality.
Changes in scores of environmental mastery as measured by Psychological well-being scale (PWB) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The Psychological Well-Being Scale is a self-report measure of eudaimonic well-being evaluated through six dimensions: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. In this trial, we will evaluate only environmental mastery. Participants respond using a six-point format: strongly disagree (1), moderately disagree (2), slightly disagree (3), slightly agree (4), moderately agree (5), strongly agree (6). Responses to negatively scored items are reversed in the final scoring procedures so that high scores indicate high self-ratings on the dimension assessed.
Change in Dispositional Optimism as measured by Life Orientation Test-Revised (LOT-R). | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  LOT-R (Scheier, Carver & Bridges, 1994) is a 10-item measure of dispositional optimism as a single bipolar dimension. Of the 10 items, 3 items measure optimism, 3 items measure pessimism, and 4 items serve as fillers. Respondents rate each item on a 4-point scale: 0 = strongly disagree, 1 = disagree, 2 = neutral, 3 =agree, and 4 = strongly agree. Scoring of the scale is based on summing the items that measure optimism and the (reverse scored) items that measure pessimism (score range 0-30 with higher values reflecting greater optimism and lower values reflecting higher pessimism).
Change in resilience as measured by Connor-Davidson ResIlience SCale (CD-RISC 10-item version). | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The CD-RISC 10 (Campbell-Sills& Stein, 2007) is a self-report measure of resilience. The 10 item version (score range 0-40, with higher scores reflecting greater resilience) comprises items 1, 4, 6, 7, 8, 11, 14, 16, 17, 19 from the original scale, and was developed by Drs. Campbell-Sills and Stein, at the University of California, San Diego, on the basis of factor analysis.
Changes in affect as measured by Positive-Negative Affect Schedule (PANAS) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  The PANAS (Watson et al, 1988) is a self-report questionnaire. The list is split up into two segments, or mood scales. One scale measures a person's positive emotion and the other scale measures the negative. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent agrees that this applies to him. The final score of the PANAS Scale / Positive and Negative Affect Schedule (PANAS) test is the sum of the 10 terms on the positive scale and the sum of the 10 terms on the negative scale. The value assigned is positive for answers on the positive scale and negative for answers on the negative scale.
Maintenance or improvement of Aerobic Capacity and Gait using 6' Minute Walking Test (6MWT) | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  6' Minute Walking Test (6MWT) is has been validated as a general indicator of overall physical performance and mobility for older people (Duncan et al 1993, Harad et al 1999). The total distance walked is measured. The Rating of Perceived Exertion will be also recorded to gain additional information.
Changes in Balance, Functional Mobility and Strength measured by 30 Second Sit to Stand Test only CHF | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  It is a measure of performance. To test functional lower limb strength and dynamic balance through repeated sit-to-stand activity. Scoring: record the number of complete stands performed in 30 seconds. Use of arms to push off or incomplete stands do not count. If a patient cannot stand even once then the score for the test is zero.
Change in motor functionality as measured by Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part-III only in Parkinson's Disease group | Baseline, post treatment (up to 3 or 4 months) and follow-up (up to 3 or 4 months)
  MDS-UPDRS part-III (Goetz et al., 2008) with 27 items. Performance measure. Administered by the clinician. Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The total UPDRS score ranging from 0-108 in which zero is the best and 100 the worst possible disability.
Change in executive functions as measured by Picture Interpretation test 360 (PIT360) only in Parkinson's disease group. | Baseline, post treatment (up to 3 or 4 months)
  Picture Interpretation test 360 (Serino et al, 2017) Scoring: Time to correct identification of the scene, with range 0-180 seconds Higher values represent a worse outcome.
Change in general cognitive function as measured by the Montreal Cognitive Assessment (MoCA) test only in Parkinson's disease group. | Baseline, post treatment (up to 3 or 4 months)
  The Montreal Cognitive Assessment (MoCA) total score ranging from 0 to 30. Higher values represent a worse outcome.
Maintaining cardiovascular performance as measured by echocardiography | Baseline, post treatment (up to 3 or 4 months)
  measure of Ejection Fraction using echocardiography as surrogate markers
Maintaining the Forced expiratory volume in the 1st second (FEV1%) as measured by spirometry (only in COPD patients) | Baseline, post treatment (up to 3 or 4 months)
  the measure of FEV1% using spirometry as surrogate marker

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Baglio, MD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi ONLUS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided